CLINICAL TRIAL: NCT05186441
Title: The Effect of Theta Burst Stimulation on the Inhibition Control Function of Bulimia Nervosa and Relevant Mechanism Study
Brief Title: The Effect of iTBS on the Inhibition Control Function of BN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Sufang PENG, attending doctor of Psychosomatic Department in Shanghai Mental Health, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20210712-SFPeng-YChen
Record Dates: First submitted 2021-08-06; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Feeding and Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DMPFC iTBS (Active Comparator): DMPFC iTBS group has 30 patients. Each receive 20 times DMPFC iTBS therapy. During the iTBS, a 5-min train treatment(110%RMT, 2s on and 8s off, 900 pulses in total）was applied to the left DMPFC.
  Interventions: Other: DMPFC iTBS
- DLPFC iTBS (Active Comparator): DLPFC iTBS group has 30 patients. Each receive 20 times DMPFC iTBS therapy. During the iTBS, a 5-min train treatment(110%RMT, 2s on and 8s off, 900 pulses in total）was applied to the left DMPFC.
  Interventions: Other: DLPFC iTBS
- placebo (Sham Comparator): The placebo research received similar pseudo-stimulation treatment, which was the same as the treatment site and method of true stimulation, but during stimulation, the coil used B65 8 zigzag coil, which was flipped 180 degrees, and only produced stimulation sound during treatment, but did not produce irritating magnetic field. It can produce a placebo effect.
  Interventions: Other: DMPFC iTBS; Other: DLPFC iTBS

INTERVENTIONS:
Other: DMPFC iTBS — The intermittent theta-burst stimulation (iTBS) (i.e. two excitatory intervention paradigm) to target DMFPC can improve out-of-control behavior and decision-making model.
  Arms: DMPFC iTBS; placebo
Other: DLPFC iTBS — The intermittent theta-burst stimulation (iTBS) to target DLFPC (i.e. region within the executive control network) can effectively reduce craving, which is probably associated with enhancement of executive function.
  Arms: DLPFC iTBS; placebo

SUMMARY:
Pathological out-of-control behavior is the core clinical symptom of Bulimia nervosa (BN). The study of its neural circuits and biological mechanism is very important to explore new intervention targets. Previous studies have found that the patients with BN have inhibitory control impairment, which may be the basis of uncontrolled binge eating and purging behaviors of BN. The study found that the cognitive decision-making dysfunction of substance addicts may lead to behavior solidification. At present, there is no related research on the cognitive decision-making model of BN. Previous studies of applicants have found that there is an enhancement in goal-oriented decision-making in BN, which may explain the binge eating and purging behaviors aimed at weight control. In addition, BN patients have obvious impulsiveness, and the individuals of BN often feel unable to control eating behavior , and experience obvious sense of out of control. The previous study confirmed that untreated BN patients were highly impulsive and had inhibitory control disorders. Inhibition and control disorder is one of the important pathogenesis of BN. Previous studies indicated that dorsolateral prefrontal cortex (DLPFC) and dorsomedial prefrontal cortex (DMPFC) were associated with aboved symptoms. In this study, the patients with BN were selected as subjects. A randomized, single-blind cohort study was designed to observe the effect of iTBS intervention of DLPFC or DMPFC on pathological out-of-control behavior. Combined with behavioral, neuroimaging and genetic techniques, the investigators focused on the function of the prefrontal lobe-striatum neural circuits dopamine system. By the objective markers of peripheral, brain imaging and behavior of BN, to provide new targets and ideas for the treatment of BN.

DETAILED DESCRIPTION:
Bulimia nervosa(BN) is a chronic and refractory mental disorder characteristic of recurrent binge eating and weight control which mostly occur in adolescents and young women. The life-time prevalence ranges from 1.0%-4.2%, and keep increasing. Pathological out-of-control behavior is the core clinical symptom of BN. Impulsive personality trait is an important risk factor for overeating symptoms in patients with BN. Inhibition control dysfunction leads to increased impulsiveness, while impaired goal-oriented control leads to rigid behavior habits, such as obsessive-compulsive drug-seeking and drug use, resulting in pathological out-of-control behavior.

Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive, safe and non-invasive physical intervention and nerve stimulation, which can be targeted at specific brain regions or networks, providing hope for people who do not respond well to drug therapy. iTBS stimulation mode can induce long-term potentiation of behavior and neural activity (LTP). Previous studies indicated that dorsolateral prefrontal cortex (DLPFC) and dorsomedial prefrontal cortex (DMPFC) were associated with out-of-control behavior.

In this study, the investigators will recruit 90 BN patients, would randomly divided into 30 DMPFC iTBS intervention group, 30 DLPFC iTBS and 30 sham-stimulation group. 20 iTBS will be given in the intervention group at DMPFC or DLPFC. To assess the eating disorder symptoms, impulsive and emotional change, clinical symptom scales, psychological scales and the behavioral experiments will be used at baseline, 4 weeks, 8 weeks, 12 weeks and16weeks, respectively. Furthermore, brain MRI will be used for BN at baseline.

This study is innovative and feasible. If the expected results can be obtained, it will lay a foundation for understanding the common mechanism behind the pathological behavior of BN and provide new directions and ideas for the design of effective intervention measures.

ELIGIBILITY:
Inclusion Criteria:

* female,
* Han nationality;
* right-handed;
* meet the diagnostic criteria of DSM-5 bulimia nervosa, body mass index (BMI) ≥ 18.5kg / m2;
* education level of junior high school or above, sufficient audiovisual level to complete the necessary examination of the study.
* Before entering the group, he has received fluoxetine treatment, the dose has been stable for one month, and has not received any form of physiotherapy (such as electroconvulsive therapy) within one month;
* each patient must understand the nature of this study and sign an informed consent form.

Exclusion Criteria:

* Patients who meet the diagnosis of DSM-5 other than BN, such as substance abuse / dependence, bipolar disorder, high risk of suicide, strong destructive impulses or antisocial behaviors;
* complicated with severe organic diseases and cognitive impairment, make it impossible for patients to complete the required symptom assessment and psychological tests;
* have a history of brain trauma or brain disease, epilepsy, etc. Those who have been exposed to ECT or MECT within 1 month;
* those with intracranial metal materials or pacemakers, implanted metal objects in vivo;
* those who are pregnant or planned pregnancy, women of childbearing age who are positive in pregnancy test.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Eating Disorder Examination(EDE-Q) | Change from Baseline eating attitudes and behaviors at 4 weeks,8weeks,12weeks,16weeks.
  EDE-Q can evaluate the eating disorder behavior and psychology characteristics and assess their frequency and intensity, which can assess the severity of eating disorders. The scores of the subscales are obtained by calculating the average of the items that comprise each subscale, and the global score (EDE-Q 6.0) is the average of scores of the four subscales. The higher is the score, the more severe in the ED-symptoms.

SECONDARY OUTCOMES:
Barratt Impulsiveness Scale(BIS-II) | Change from Baseline the severity of impulse suppression orientation at 4 weeks,8weeks,12weeks,16weeks.
  This tool can measure the severity of impulse suppression orientation.The total score for BIS-11 ranges from 30 to 120. The higher is the score, the higher is the impulsiveness.
Beck Depression Inventory-II (BDI- II) | Change from Baseline the severity of the symptoms of depression at 4 weeks,8weeks,12weeks,16weeks.
  Depression symptoms were assessed with the BDI-II. The scale has 21-items. The total score for BDI- IIranges from 0 to 84.The higher is the score, the higher is the depression.
Beck Anxiety Inventory (BAI) | Change from Baseline Baseline the severity of the symptoms of anxiety at 4 weeks,8weeks,12weeks,16weeks.
  BAI is a 21-item self-report scale for assessing the symptom of anxiety. The total score for BAI ranges from 0 to 84. The higher is the score, the higher is the anxiety.
Behavioral experiment(Sequential learning task ) | Change from Baseline behaviors at 4 weeks.
  The spaceship task from Decker et al will be used. The task was designed to dissociate model-free and model-based learning strategies. The goal of the participants will to collect "space gems". In the first stage, the participants choose between two spaceships. The probability of each spaceship's transition to two planets is fixed. In the second stage, on each planet, participants need to choose between two aliens to obtain gems. The probability of getting a gem changes slowly at this stage. This changing reward probability encourages participants to explore different options throughout the task to maximize the reward. The behavior data will be modeled, and the hybrid reinforcement learning model will used to obtain the ratio of model-based behavior and model-free behavior in the process of individual learning decision-making.
Incidence of Adverse Events [Safety and Tolerability] (i.e., seizures, etc.) | through study completion, an average within 1 week
  The frequency of adverse events from each participant.
Behavioral experiment(Stop-signal task ) | Change from Baseline behaviors at 4 weeks.
  The stop-signal task was adjusted using as cues the two foods previously selected after the rating session. Two types of conditions were included, such as low-error condition and high-error condition. Participants performed 240 trials in total: 160 Go trials (80 for the Low-Error condition and 80 for the High-Error condition) and 80 Stop trials (40 for the Low-Error condition and 40 for the High-Error condition). The task lasted approximately 16 minutes. Data analysis will be performed on the accuracy (number of errors) and the RTs of correct responses vs. errors (no-response trials ignored), for the Low- vs. High-Error condition, and for Go vs. Stop trials.
Behavioral experiment(Delay discounting task ) | Change from Baseline behaviors at 4 weeks.
  The delay discounting task for monetary present choices between differing amounts of reward at varing time points (such as 2 days, 7days, 15days, 1 month, 45 days, 3 months, 6 months and 1 year), where one of the options is a smaller amount of reward available soon or immediately, and the other option is a larger amount of reward available after a longer delay. Discount rate will be estimated by fitting the indifference point data to a discounting model.
MRI | before the intervention
  brain activation and structure as assessed by MRI

CONTACTS AND LOCATIONS:
Overall Officials: SuFang Peng, PhD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China